CLINICAL TRIAL: NCT02707926
Title: The Lymphoid Tissue Pharmacology of Antiretroviral Drugs
Status: Withdrawn | Type: Observational
Why Stopped: COVID-19 required halting recruitment into new clinical protocols. Following the allowed opening to clinical research, our assessment of site and investigator interest and time frame of available grant funding resulted in a judgment of futility.
Sponsor: University of Nebraska (Other)
Collaborators: University of Minnesota (Other); National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Responsible Party: Sponsor
Other Study IDs: 0212-16-ET; 1R01AI124965-01 (NIH)
Record Dates: First submitted 2016-03-03; First posted 2016-03-14 (Estimated); Last update posted 2023-08-24 (Actual); Status verified 2023-08

CONDITIONS: HIV Infection
MeSH Terms: conditions — HIV Infections | interventions — Anti-HIV Agents; Anti-Retroviral Agents

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Blood, urine, lymph node biopsy, colonoscopy biopsy of ileum and rectum
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: Anti-HIV Agents — Therapy to treat HIV infection
  Other Names: antiretroviral (ARV) HIV drugs

SUMMARY:
Hypothesis:

Antiretroviral drugs (ARVs) with enhanced LT penetration characteristics in vitro and in macaques will translate into an ARV regimen with increased LN and GALT concentrations and a faster decay and more potent suppression of HIV replication in LT in HIV-infected persons.

Objectives:

1. Determine lymph nodes (LN) and gut-associated lymphoid tissue (GALT) pharmacokinetics (PK) in HIV-infected persons on an antiretroviral drug (ARV) regimen.
2. Determine virological responses of antiretroviral therapy in plasma, peripheral blood mononuclear cells (PBMCs) and lymphoid tissue (LT).

DETAILED DESCRIPTION:
This is a single-center study of 18 ARV naïve, HIV infected persons to assess impact of an ARV regimen on lymph node (LN) and (GALT) virus reservoirs.

All participants will give informed consent. At baseline, plasma and PBMCs will be obtained and all subjects will have an incisional biopsy of an inguinal LN and pinch biopsy of ileum and rectum via colonoscopy. The selected LT-enhanced ARV regimen will be initiated. Participants will return to the clinic at weeks 2 and 4 and then monthly for safety evaluations, CD4 T cell counts, plasma HIV-RNA and ARV drug concentrations in plasma and PBMCs. An intensive PK study will be performed at week 2. At months 3 and 6, the inguinal LN biopsy and pinch biopsies of ileum and rectum will be repeated.

ELIGIBILITY:
Inclusion Criteria:

1. Antiretroviral drug (ARV)-naive, HIV-infected individuals
2. Aged 18 years or over
3. Agree to initiating ARV therapy
4. BMI ≤ 30
5. Inguinal lymph node(s) identifiable by ultrasound at enrollment
6. Screening plasma HIV RNA > 40,000 copies/mL
7. Screening CD4 count > 200 cells/mm3
8. Women of child bearing potential must agree to use effective contraception while on the study.
9. Screening viral isolates demonstrate genotype sensitivity to chosen antiretroviral therapy (ART) regimen.
10. Able to provide voluntary written consent

Exclusion Criteria:

1. Previous ARV therapy
2. Contraindications to ARV regimen (e.g., comorbid conditions or drug interactions), or study procedures as determined by the principal investigator.
3. Planning or current pregnancy or breastfeeding
4. History and/or presence of any clinically significant disease or disorder, such as cardiovascular, pulmonary, renal, hepatic, neurological, gastrointestinal and psychiatric/mental disease/disorder, which, in the opinion of the enrolling physician, may put the participant at risk because of participation in the study, influence the results of the study, or affect the participant's ability to participate in the study.
5. Inability to comply with study procedures per enrolling physician discretion

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Eighteen (18) antiretroviral drug (ARV)-naive, HIV-infected persons who are going to initiate ARV therapy will be recruited at the University of Minnesota. Study entry is open to adults regardless of race or ethnic background. While there will be every effort to seek out and include minority participants from both genders, the patient population is expected to be no different than that of the HIV infected population in Minnesota.
Sampling Method: Non-Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2023-03-25 (Actual); Primary Completion 2023-08-17 (Actual); Study Completion 2023-08-17 (Actual)

PRIMARY OUTCOMES:
Lymph node (LN) tissue penetration ratio. | 6 months
  Ratio of antiretroviral drug concentration in lymph node (LN) to peripheral blood mononuclear cells (PBMCs)
Lymph node (LN) residual viremia. | 6 months
  Quantification of residual viremia in lymph node (LN) at 6 months of therapy as measured by digital droplet polymerase chain reaction (PCR), which can quantify as low as 50 copies/million cells.

CONTACTS AND LOCATIONS:
Overall Officials: Tim Schacker, MD, Principal Investigator — University of Minnesota; Courtney V Fletcher, PharmD, Principal Investigator — University of Nebraska

IPD SHARING:
Plan to Share IPD: Yes
The results of this trial will be of interest to the HIV research and medical communities. We expect to submit the data from the main analysis within 6 months of completing the work. We will publish the results in a major scientific journal and present the results at a major scientific meeting (e.g., CROI). Subsequent analyses will be presented at national and international HIV meetings. Data generated under this project, and any intellectual property, will be administered in accordance with NIH policies, including the NIH Data Sharing Policy the NIH Public Access Policy.
Time Frame: 6 months of completing the work
Access Criteria: Data generated under this project, and any intellectual property, will be administered in accordance with NIH policies, including the NIH Data Sharing Policy the NIH Public Access Policy.

REFERENCES:
- [Background] Lorenzo-Redondo R, Fryer HR, Bedford T, Kim EY, Archer J, Pond SLK, Chung YS, Penugonda S, Chipman J, Fletcher CV, Schacker TW, Malim MH, Rambaut A, Haase AT, McLean AR, Wolinsky SM. Persistent HIV-1 replication maintains the tissue reservoir during therapy. Nature. 2016 Feb 4;530(7588):51-56. doi: 10.1038/nature16933. Epub 2016 Jan 27. PMID 26814962
- [Background] Fletcher CV, Staskus K, Wietgrefe SW, Rothenberger M, Reilly C, Chipman JG, Beilman GJ, Khoruts A, Thorkelson A, Schmidt TE, Anderson J, Perkey K, Stevenson M, Perelson AS, Douek DC, Haase AT, Schacker TW. Persistent HIV-1 replication is associated with lower antiretroviral drug concentrations in lymphatic tissues. Proc Natl Acad Sci U S A. 2014 Feb 11;111(6):2307-12. doi: 10.1073/pnas.1318249111. Epub 2014 Jan 27. PMID 24469825